CLINICAL TRIAL: NCT04128371
Title: Pilot Study of Mepolizumab in Episodic Angioedema With Eosinophilia
Brief Title: Mepolizumab in Episodic Angioedema With Eosinophilia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was closed after the first five participants completed their participation due to lack of efficacy.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200002; 20-I-0002
Record Dates: First submitted 2019-10-15; First posted 2019-10-16 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2022-11

CONDITIONS: Eosinophilia; Angioedema
Keywords: Absolute Neutrophil Count; Cycling; Gleich's Syndrome; Urticaria; Serum Interleukin 5
MeSH Terms: conditions — Eosinophilia; Angioedema; Urticaria | interventions — mepolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active treatment (Experimental): Participants with episodic angioedema with eosinophilia (EAE) received mepolizumab 700 mg intravenously monthly for three doses.
  Interventions: Biological: mepolizumab

INTERVENTIONS:
Biological: mepolizumab — Mepolizumab is a fully humanized monoclonal antibody (IgG1, kappa mAb) supplied as 100 mg of lyophilized powder in sterile, single-dose vials. Mepolizumab 100 mg vials were reconstituted according to the manufacturer, for a total dose of 700mg administered as intravenous infusion.
  Other Names: Nucala

SUMMARY:
Background:

Gleich syndrome is also called episodic angioedema with eosinophilia (EAE). People with EAE have episodes of swelling. They may also have itching, hives, fever, and weight gain. During episodes, the body has very high numbers of white blood cells, especially a kind called eosinophils. Researchers think a drug called mepolizumab could help.

Objective:

To see if mepolizumab causes EAE symptoms to be less severe and happen less often.

Eligibility:

People ages 18 or older with EAE.

Design:

Participants will be screened under NIH protocol 94-I-0079.

Participants will have 8 visits over about 6 months. The timing of some visits will depend on each participant s EAE episodes. Visits will include:

* Medical history
* Physical exam
* Blood and urine tests
* Optional bone marrow collection at first or second visit. For this, a needle will be inserted through the participant s hip bone into the marrow.

Participants will get mepolizumab 3 times over about 3 months. They will get their first dose when their eosinophils are at their lowest point. They will get the drug by IV. A needle will guide a thin plastic tube into an arm vein. The drug will be given through the tube over about 30 minutes.

Participants will keep a daily online log for about 3 months. The log will track their weight, temperature, and EAE symptoms. During the whole study, they will complete 2 online questionnaires about their symptoms. They will fill out 1 daily and 1 monthly.

Participants will have blood and urine tests 2-3 times a week. For these, they will go to their local doctor.

DETAILED DESCRIPTION:
Episodic angioedema with eosinophilia (EAE), also known as Gleich s Syndrome,is a rare disorder characterized by recurrent episodes of urticaria, fever, angioedema, weight gain and dramatic eosinophilia that occur at 3- to 6-week intervals and resolve with spontaneous diuresis in the absence of therapy. Although the syndrome is often classified in the broad category of idiopathic hypereosinophilic syndrome (HES), EAE is a distinct eosinophilic syndrome that is remarkably homogeneous in clinical presentation. More recently, it has become apparent that there is multilineage cycling, involving lymphocytes and neutrophils in addition to eosinophils. Early studies described cyclic elevations of serum interleukin 5 (IL-5) preceding the rise in eosinophilia, and additional studies have shown cyclic elevations in other type II cytokines as well as in eosinophilic chemokines. Aberrant T cells with a CD3-CD4+ surface phenotype have also been detected in the majority of subjects with EAE. The cyclic nature of the disorder and the involvement of multiple cell lineages have made it difficult to determine the underlying cause of EAE.

We hypothesize that IL-5 driven eosinophilia is central to the pathogenesis of EAE. Suppression of eosinophil cycling by blocking IL-5 would help determine whether eosinophils are indeed the main drivers of the symptoms of angioedema and urticaria and pave the way for future mechanistic studies investigating the etiology of this unusual disorder. The purpose of this pilot study is to evaluate the effect of mepolizumab, a humanized antibody to IL-5, on eosinophil cycling in 12 subjects with EAE. Subjects with EAE will undergo screening on the National Institutes of Health protocol 94-I-0079 to establish the periodicity of their cycling (if not previously determined) and the optimal timing for the baseline visit. After screening, subjects will be followed closely with signs and symptoms recorded in a daily log and daily and monthly questionnaires, as well as complete blood counts and research blood collected for one cycle prior to administration of mepolizumab. Subjects will receive a total of 3 monthly administrations of mepolizumab at 700 mg, followed by drug de-escalation over 6 additional monthly administrations for subjects who demonstrate benefit from mepolizumab. All subjects will have a follow-up visit about 1 month after the last study administration of mepolizumab.

The primary efficacy endpoint will be reduction of symptoms and severity of symptoms after mepolizumab. Secondary endpoints will include reduction in peak eosinophils after mepolizumab, continued suppression of absolute eosinophil count and reduction in symptoms following monthly dosing of mepolizumab therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:

A subject will be eligible for participation in the study only if all of the following criteria apply:

1. The subject is male or female, aged 18 years or older.
2. The subject has a documented diagnosis of EAE.
3. The subject has symptoms of EAE in the cycle prior to screening, including but not limited to fever, swelling, hives or rashes, weight gain, muscle pain, and lymphadenopathy.
4. Cycling of eosinophils is ongoing as indicated by a peak absolute eosinophil count (AEC) greater than or equal to 1500/mm^3 during at least one cycle in the prior 3 months.
5. If taking corticosteroids, the subject is able and willing to stay on a stable dose for 6 weeks prior to screening.
6. The subject agrees to storage of study samples.
7. The subject is able to provide informed consent.
8. Females are eligible for this study if they are:

   * of non-childbearing potential (i.e., women who have had a hysterectomy or tubal ligation or are postmenopausal as defined by no menses in 1 year); OR
   * of childbearing potential but willing to practice effective contraception or abstinence during administration of the study drug and for 100 days (5 terminal half-lives) after administration of the study drug.
   * Not breastfeeding.

Participation of Women:

Pregnancy: The effects of mepolizumab on the developing human fetus are unknown. For this reason, women of childbearing potential must agree to use adequate contraception (see below for acceptable methods) prior to study entry, for the duration of study participation, and for >5 terminal half-lives (approximately 100 days) after administration of the last dose of study drug. Nonreproductive potential is defined as post-menopausal, male partner who has azoospermia or is surgically sterile (at least 6 weeks before screening) and is the sole sexual partner, surgical sterility, or a congenital or acquired condition that definitely prevents conception. Further, postmenopausal is defined as at least 12 consecutive months with no menses at age 50 or older, or a high follicle-stimulating hormone level in the postmenopausal range at ages 45-50 years in subjects not using hormonal contraception or hormone replacement therapy.

Females with reproductive potential must either practice complete and uninterrupted abstinence from heterosexual activity or use 2 of the following methods of contraception with their partners. The 2 methods must include either 2 barrier methods, or 1 barrier method and 1 non-barrier method, both of which must be consistently used:

Barrier Methods:

1. Diaphragm with spermicide
2. Cervical cap with spermicide or contraceptive sponge (for nulliparous subjects only)
3. Male or female condom (cannot be used together)

Non-Barrier Methods

1. An intrauterine device with a documented failure rate of <1%
2. Hormonal contraception: pill (estrogen/progestin or progestin-only), patch, vaginal ring, rod implanted in the skin, or subcutaneous injection methods

Females of childbearing-potential must have a negative pregnancy test result prior to receiving mepolizumab at each on-site study visit. During the course of the study, if a woman becomes pregnant or suspects she is pregnant, she should inform the study staff and her primary care physician immediately. A pregnancy registry has been created for subjects who become pregnant while receiving the approved dose of mepolizumab (100 mg subcutaneous injection) for asthma.

Fertility: There is no fertility data in humans. Animal studies showed no adverse effects of anti-IL-5 treatment on fertility.

EXCLUSION CRITERIA:

A subject will not be eligible to participate in the study if any of the following conditions are fulfilled at the time of screening:

1. Treatment with immunosuppressive or immunomodulatory agents including but not limited to cyclosporine, interferon-alpha, azathioprine, methotrexate, and cyclophosphamide within the past 3 months.
2. Treatment with biologics including but not limited to mepolizumab, IVIG, anti-TNF agents, rituximab, benralizumab, alemtuzumab, reslizumab, dupilumab, lebrikizumab, and omalizumab within 6 months or 5 half-lives (whichever is longer). Subjects who received rituximab at any time in the past must have normal B-cell numbers to participate.
3. Co-morbid illness, alcohol or substance abuse, or any other condition (e.g., HIV, active hepatitis) that, in the opinion of the investigator, places the subject at undue risk by participating in the study.
4. Treatment with a daily dose of corticosteroids >40 mg.

Co-enrollment Guidelines: Co-enrollment in other trials is restricted, other than enrollment on observational studies or those evaluating the use of a licensed medication. Study staff should be notified of co-enrollment as it may require the approval of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paneez Khoury, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Rothenberg ME, Klion AD, Roufosse FE, Kahn JE, Weller PF, Simon HU, Schwartz LB, Rosenwasser LJ, Ring J, Griffin EF, Haig AE, Frewer PI, Parkin JM, Gleich GJ; Mepolizumab HES Study Group. Treatment of patients with the hypereosinophilic syndrome with mepolizumab. N Engl J Med. 2008 Mar 20;358(12):1215-28. doi: 10.1056/NEJMoa070812. Epub 2008 Mar 16. PMID 18344568
- [Background] Gleich GJ, Schroeter AL, Marcoux JP, Sachs MI, O'Connell EJ, Kohler PF. Episodic angioedema associated with eosinophilia. N Engl J Med. 1984 Jun 21;310(25):1621-6. doi: 10.1056/NEJM198406213102501. PMID 6727934
- [Background] Khoury P, Herold J, Alpaugh A, Dinerman E, Holland-Thomas N, Stoddard J, Gurprasad S, Maric I, Simakova O, Schwartz LB, Fong J, Lee CC, Xi L, Wang Z, Raffeld M, Klion AD. Episodic angioedema with eosinophilia (Gleich syndrome) is a multilineage cell cycling disorder. Haematologica. 2015 Mar;100(3):300-7. doi: 10.3324/haematol.2013.091264. Epub 2014 Dec 19. PMID 25527564
- [Result] Khoury P, Makiya MA, Rahim R, Bowman A, Espinoza D, Schiffenbauer A, Koch M, Anderson C, Constantine G, Maric I, Sun X, Pittaluga S, Brown T, Ware JM, Wetzler L, Fay MP, Klion AD. Mepolizumab incompletely suppresses clinical flares in a pilot study of episodic angioedema with eosinophilia. J Allergy Clin Immunol. 2024 Mar;153(3):821-830.e6. doi: 10.1016/j.jaci.2023.11.002. Epub 2023 Nov 10. PMID 37951310
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-I-0002.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Treatment
Started | 5
Completed | 4
Not Completed | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Active Treatment
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Maximum Daily Angioedema Activity Score (AAS)
Description: We measure the number and severity of clinical symptoms associated with episodic angioedema with eosinophilia (EAE) using the maximum of the patient reported daily angioedema activity score, a validated patient reported outcome measure. The daily score was used to measure changes in swelling within a cycle. Participants answered 5 questions each day that were scored from 0-3 for each item. The daily score consisted of a minimum score of 0 and a maximum score of 15, the sum of the 5 question answers. Higher scores indicate a worse outcome. The change of the daily angioedema activity score is measured as the average percent reduction in the maximum score over the 3 cycles (about 3 months) after treatment compared to the cycle (about 1 month) pre-treatment. The estimated percent change and its confidence interval was calculated from a quasi-Poisson model. The model estimates a multiplicative treatment effect on the baseline AAS, and that effect is translated into a percent change.
Time Frame: 1 month prior to treatment and 3 months after treatment
Population: The analyses included all participants during the cycle (about the 1 month) prior to treatment with up to 3 cycles (about 3 months) after treatment began. One patient withdrew after only 2 cycles post treatment and we used their values up until time of withdrawal.
Measure: Number (95% Confidence Interval); unit: Percent change
Arm/Group | Active Treatment
Number analyzed (Participants) | 5
Percent change | 16.5 [-64.6 to 57.7]

2. Secondary Outcome: Percent Change in Peak Absolute Eosinophil Count (AEC)
Description: Percent change in peak AEC is measured on each individual as the percentage change in peak AEC in the cycle following the first mepolizumab infusion compared to the peak AEC in the cycle prior to mepolizumab treatment. Those values are summarized by taking the mean of a transformation of each percent change in peak AEC, and back-transforming the results. Specifically, if x is the percent change in peak AEC, then the transformation is log(1-x/100). The estimated percent change and its confidence interval was calculated using the mean of the transformed values and using the associated one-sample t-test confidence interval on that mean, then translating those estimates and confidence intervals back to the percent change scale.
Time Frame: 1 month prior to treatment and 1 month after treatment
Population: Analysis included all participants
Measure: Number (95% Confidence Interval); unit: Percent change
Arm/Group | Active Treatment
Number analyzed (Participants) | 5
Percent change | 82.2 [-108.5 to 98.5]

3. Secondary Outcome: Percent Change in Peak Absolute Eosinophil Count (AEC)
Description: Percent change in peak AEC is measured on each individual as the percentage change in peak AEC by visit 8 (3 months) compared to the peak AEC in the cycle prior to mepolizumab treatment. Those values are summarized by taking the mean of a transformation of each percent change in peak AEC, and back-transforming the results. Specifically, if x is the percent change in peak AEC, then the transformation is log(1-x/100). The estimated percent change and its confidence interval was calculated using the mean of the transformed values and using the associated one-sample t-test confidence interval on that mean, then translating those estimates and confidence intervals back to the percent change scale.
Time Frame: 1 month prior to treatment and 3 months after treatment
Population: 4 of the 5 participants were assessed at visit 8. One participant withdrew prior to visit 8, and we used their values at visit 7.
Measure: Number (95% Confidence Interval); unit: Percent change
Arm/Group | Active Treatment
Number analyzed (Participants) | 5
Percent change | 96.2 [71.4 to 99.5]

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | Active Treatment
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Treatment (N=5)
Nausea (Gastrointestinal disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Coronavirus test positive (Investigations) | 2
Haemoglobin decreased (Investigations) | 1
Paraesthesia (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
Study was closed due to futility

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/71/NCT04128371/Prot_SAP_000.pdf